CLINICAL TRIAL: NCT07249814
Title: Comparison of Fractionated Versus Bolus Administration of Different Doses of Hyperbaric Bupivacaine Combined With Opioids in Spinal Anesthesia for Caesarean Section - A Prospective, Randomized, Single Blind Clinical Trial
Brief Title: Comparison of Fractionated Versus Bolus Administration of Different Doses of Hyperbaric Bupivacaine Combined With Opioids in Spinal Anesthesia for Caesarean Section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bogomolets National Medical University (Other)
Responsible Party: Principal Investigator, Kateryna Bielka, Prof., Bogomolets National Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 196
Record Dates: First submitted 2025-11-14; First posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Spinal Anesthesia for Cesarean Section
Keywords: Spinal Anesthesia; Hypotension; Hemodynamic Stability; Bupivacaine; Bolus Dose; Fractionated Dose; Cesarean Section
MeSH Terms: conditions — Hypotension

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Bolus bupivacaine (0.07 mg/cm) (Active Comparator)
  Interventions: Procedure: Bolus anesthesia
- Fractionated bupivacaine (0.07 mg/cm) (Experimental)
  Interventions: Procedure: Fractionated anesthesia
- Fractionated bupivacaine (0.06 mg/cm) (Active Comparator)
  Interventions: Procedure: Fractionated anesthesia

INTERVENTIONS:
Procedure: Fractionated anesthesia — * Group F7: received a fractionated administration of bupivacaine (0.07 mg/cm);
  * Group F6: received a fractionated administration of the reduced dose of bupivacaine (0.06 mg/cm).
  Arms: Fractionated bupivacaine (0.06 mg/cm); Fractionated bupivacaine (0.07 mg/cm)
Procedure: Bolus anesthesia — • Group B: received a bolus administration of the total dose of 0.5% hyperbaric bupivacaine (0.07 mg/cm height)
  Arms: Bolus bupivacaine (0.07 mg/cm)

SUMMARY:
This study aimed to compare the effectiveness and safety of fractionated versus bolus administration of different doses of hyperbaric bupivacaine (0.06 and 0.07 mg/cm height) combined with opioids in spinal anesthesia for cesarean section, with detailed evaluation of maternal hemodynamic effects, block characteristics and side effects.

ELIGIBILITY:
Inclusion Criteria:

* singleton full-term pregnancy scheduled for cesarean section under spinal anesthesia
* ASA physical status II-III
* age 18-50 years
* height from 140 to 180 cm
* body weight from 40 to 130 kg

Exclusion Criteria:

* patient refusal
* contraindications to spinal anesthesia
* allergy to amide-type local anesthetics

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 99 (Actual)
Dates: Start 2024-06-30 (Actual); Primary Completion 2025-06-15 (Actual); Study Completion 2025-06-15 (Actual)

PRIMARY OUTCOMES:
Hemodynamic Stability (systolic, diastolic and mean arterial pressure, heart rate) | Perioperative/Periprocedural - before spinal anesthesia and then during the cesarean section until its completion
  Hemodynamic parameters were recorded every 2 minutes for 10 minutes, then every 5 minutes until 30 minutes, then every 15 minutes until surgery completion.

SECONDARY OUTCOMES:
Spinal block characteristics (sensory block level and duration, motor block duration, analgesia duration) | Perioperative/Periprocedural
  Spinal block characteristics were assessed every minute for 5 minutes, then every 5 minutes until peak effect, then every 30 minutes until sensory regression to L1 dermatome and motor block regression to Bromage 0.
  Sensory block was assessed using pin-prick method at the midaxillary line bilaterally. Motor block was evaluated using the modified Bromage scale (0 = full motor function, 3 = complete motor block). Postoperative pain was assessed using numeric rating scale (NRS) every 30 minutes for 2 hours, then hourly for 8 hours.

CONTACTS AND LOCATIONS:
Locations (1):
- Kyiv Perinatal Center, Kyiv, Ukraine